CLINICAL TRIAL: NCT04786353
Title: Long COVID Kids DK - Investigating Long-term Hospitalizations, GP Visits, Co-morbidities, Drug Prescriptions and Symptoms in Danish Children With Covid-19
Brief Title: Long COVID Kids DK - Investigating Long-term Covid-19
Status: Active, not recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Selina Kikkenborg Berg, Professor, Rigshospitalet, Denmark
Other Study IDs: Long COVID-19 Kids DK
Record Dates: First submitted 2021-03-01; First posted 2021-03-08 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Covid-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID positive kids: Children with at least one positive SARS-CoV-2 test.
  Interventions: Other: LongCOVIDkidsDK
- Controls: Children with no positive SARS-CoV-2 test.

INTERVENTIONS:
Other: LongCOVIDkidsDK — Exposure: To be identified as an exposure for the current study, children from 0-18 years with at least one positive SARS-CoV-2 test will be identified from COVID-19 data from January 2020 until the last updated version. To be able to identify the parents who will receive the questionnaires we will also need CPR-data on the children's parents.
  Groups: COVID positive kids

SUMMARY:
During the COVID-19 pandemic children have been perceived as a group not being especially affected, with less being infected, low symptom burden and low mortality. A small proportion however develop life-threatening hyperinflammation (mis-c) and at least one Danish child has died from this condition. Since the fall of 2020 international awareness has been raised by parents reporting that their children experience gastrointestinal issues, chest pain, headaches, fatigue, joint/muscle pain, sore throat, dizziness, nausea and fever for months following COVID-19 infection.

In this study the investigators aim to investigate the proportions of possible long covid in the 45.000 Danish children that has been tested positive for covid-19. The investigators know from the Danish Covid-19 surveillance data that 300 has been admitted to the hospital within the first 2 weeks after diagnosing. However, no knowledge about how many visits the participants have to the ER and GP compared to children without covid-19 as well as hospital admissions within the first year and medical prescriptions within the first year. This knowledge can give the investigators an indication of how affected these children are on the long term. Furthermore, data has been collected about the long-term symptoms in adults, but not children, and it now seems obvious that this data are needed to fully understand the disease and orchestra the relevant medical attention for children during the covid-19 pandemic.

DETAILED DESCRIPTION:
Objectives

WP 1 Objective: to investigate long COVID symptoms after 3,6,9 and 12 months in children tested positive for SARS-CoV-2 compared to children without a positive test.

WP 2 Objective: to describe whether there is a difference in the number of visits to general practitioner, emergency department and hospitalizations in children with and without SARS-CoV-2. In addition, which co-morbid diagnoses are given 3,6,9 and 12 months after diagnosis with COVID and which drugs are prescribed.

Methods

Design: National register study and questionnaire survey.

Outcomes

WP1: Long-term COVID-19 symptoms in children will be identified from questionnaires.

WP2: To determine the difference in number of contacts to the general practitioner, emergency departments and hospitalizations in both children with and without SARS-CoV-2, an identification from COVID-19 data linked with LPR3 and SSR will occur. Identification of co-morbidities will be identified from LPR3 and prescribed drugs are available from LMDB.

Statistical analyses

WP1: To investigate parent and child reported long COVID symptoms numbers and percentages will be presented followed by multiple logistic models offered as odds ratios (OR) with 95% confidence intervals (CI).

WP2: Multiple regressions models presented as OR with 95% CI will be used to examine the differences in contacts regarding the general practitioner, emergency departments, hospitalizations, co-morbidities and prescribed drugs in children with and without COVID.

All analyses will be stratified by age groups and gender.

Population

Exposure: To be identified as an exposure for the current study, children from 0-18 years with at least one positive SARS-CoV-2 test will be identified from COVID-19 data from January 2020 until the last updated version. To be able to identify the parents who will receive the questionnaires the investigators will also need CPR-data on the children's parents.

Non-exposure: Children from 0-18 years without a positive SARS-CoV-2 test for the entire period of January 2020 until the last updated version will be identified from the Danish Civil Registration System. To be able to identify the parents who will receive the questionnaires the investigators will need CPR-data on the parents.

Variables

COVID-19 data will enable information on children with and without positive SARS-CoV-2 tests. The parents who will receive questionnaires will also be identified from this register likewise will data on death, sex and age.

The Temporary Danish National Patient Register (LPR3) will provide data on the number of emergency visits, hospitalizations and co-morbidities.

The Danish Health Insurance Register (SSR) offers numbers of contacts with the general practitioner.

The Danish Medicines Registry (LMDB) enables the investigators to link prescribed drugs.

All registers will be updated monthly by The Danish Health Authorities and the investigators will need data extraction in the period 2020 until the last updated version from all the above-mentioned registers.

Publications of results

All results will be published in international scientist journals as well as the hospital webpage and press releases.

Perspectives

This will be the largest investigation of long COVID in children to date. Denmark has excellent registers and logistics for questionnaires providing a unique opportunity to report on children's health care seeking behavior and symptoms after being infected with COVID-19. Children are an overlooked group during the pandemic and these data will provide essential information for health care staff, politicians and parents.

ELIGIBILITY:
Inclusion Criteria:

* must be included in the covid-19 monitoring database

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Exposure: To be identified as an exposure for the current study, children from 0-18 years with at least one positive COVID-19 test will be identified from Covid-19 data from January 2020 until the last updated version. To be able to identify the parents who will receive the questionnaires we will also need CPR-data on the children's parents.
  Non-exposure: Children from 0-18 years without a positive COVID-19 test for the entire period of January 2020 until the last updated version will be identified from Covid-19 data. To be able to identify the parents who will receive the questionnaires we will need CPR-data on the parents.
Sampling Method: Non-Probability Sample
Enrollment: 330000 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Contacts to the general practitioner | Up to 1 year after diagnosis with covid-19
  To determine the difference in number of contacts to the general practitioner, in children with and without COVID-19, an identification from the Danish COVID-19 database linked with the Danish Health Insurrance Register will occur.
Hospitalizations | Up to 1 year after diagnosis with covid-19
  To determine the number of hospitalizations in children with and without COVID-19, an identification from the Danish COVID-19 database linked with the Danish National Patient Register will occur.
Diagnoses | Up to 1 year after diagnosis with covid-19
  To determine which diagnoses the children with covid-19 are given compared to children without covid-19, an identification from the Danish COVID-19 database linked with the Danish National Patient Register will occur.
Prescribed drugs | Up to 1 year after diagnosis with covid-19
  To determine which drugs the children with COVID-19 are given compared to children without covid-19, an identification from the Danish COVID-19 database linked with the Danish Medicines Registry will occur.
Long COVID symptoms | Up to 1 year after diagnosis with covid-19
  Through self-reported (by child or parent) survey data long COVID symptoms will be evaluated among children with and without COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Selina K Berg, PhD, Principal Investigator — 29190623
Locations (1):
- Rigshospitalet, Copenhagen University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bering L, Christensen AV, Birk NM, Thygesen LC, Bundgaard H, Benfield T, Nygaard U, Johannesen J, Nielsen SD, Berg SK. Risk of New-onset Type 1 Diabetes in Danish Children and Adolescents After SARS-CoV-2 Infection: A Nationwide, Matched Cohort Study. Pediatr Infect Dis J. 2023 Nov 1;42(11):999-1001. doi: 10.1097/INF.0000000000004063. Epub 2023 Aug 3. PMID 37566892
- [Derived] Kikkenborg Berg S, Palm P, Nygaard U, Bundgaard H, Petersen MNS, Rosenkilde S, Thorsted AB, Ersboll AK, Thygesen LC, Nielsen SD, Vinggaard Christensen A. Long COVID symptoms in SARS-CoV-2-positive children aged 0-14 years and matched controls in Denmark (LongCOVIDKidsDK): a national, cross-sectional study. Lancet Child Adolesc Health. 2022 Sep;6(9):614-623. doi: 10.1016/S2352-4642(22)00154-7. Epub 2022 Jun 23. PMID 35752194
- [Derived] Kikkenborg Berg S, Dam Nielsen S, Nygaard U, Bundgaard H, Palm P, Rotvig C, Vinggaard Christensen A. Long COVID symptoms in SARS-CoV-2-positive adolescents and matched controls (LongCOVIDKidsDK): a national, cross-sectional study. Lancet Child Adolesc Health. 2022 Apr;6(4):240-248. doi: 10.1016/S2352-4642(22)00004-9. Epub 2022 Feb 8. PMID 35143771